CLINICAL TRIAL: NCT02003898
Title: Post Approval Study of the TS (Threshold Suspend) Feature With a Sensor-Augmented Pump System Supplemented With Commercial Patient Data
Brief Title: Post Approval Study of the TS Feature With the 530G Pump System Supplemented With Commercial Patient Data
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP266
Record Dates: First submitted 2013-11-25; First posted 2013-12-06 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Diabetes
Keywords: Diabetes; Insulin pump; Threshold Suspend
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: All subjects are assigned to treatment with the Medtronic 530G Insulin Pump
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Medtronic MiniMed 530G Insulin Pump (Experimental): All subjects received diabetes treatment using the Medtronic MiniMed 530G insulin pump.
  Interventions: Device: Medtronic MiniMed 530G Insulin Pump

INTERVENTIONS:
Device: Medtronic MiniMed 530G Insulin Pump

SUMMARY:
The purpose of this study is to evaluate the Threshold Suspend (TS) feature of the Medtronic MiniMed® 530G insulin pump in patients 16 and older with insulin requiring diabetes.

DETAILED DESCRIPTION:
Multi-center trial is initiated to observe the Threshold Suspend (TS) feature with a sensor-augmented insulin pump (Medtronic MiniMed® 530G insulin pump) in patients 16 and older with insulin requiring diabetes over a period of one year.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is age 16 or older at time of screening
2. Subject has been diagnosed with diabetes mellitus for at least one year prior to screening.
3. Subject is currently on pump therapy.
4. Subject is transitioning to the 530G insulin pump system with the TS feature turned ON.
5. Subject is willing to complete all study related activities
6. Subject is willing to upload data every 21 days from the study pump
7. Subject must have Internet access and access to a computer system that meets the requirements for uploading the pumps. This may include use of family or friend's computer system with Internet access.
8. Subject is able (by insurance or financial means) to cover the initial investment and ongoing cost of the 530G insulin pump and consumables, CGM, Bayer CONTOUR Next Link RF enabled meter and supplies for the length of the study- 1 year.

Exclusion Criteria:

1. Subject is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study devices in the last 2 weeks.
2. Subject is a woman of child-bearing potential who has a positive pregnancy test at screening or plans to become pregnant during the course of the study
3. Subject is being treated for hyperthyroidism at time of screening
4. Subject has an abnormality (>1.8mg/dL) in creatinine at time of screening visit
5. Subject has an abnormality (out of reference range) in thyroid-stimulating hormone (TSH) at time of screening visit. If TSH is out of range, Free T3 and Free T4 will be tested. Subject may be included with TSH out of range as long as Free T3 and Free T4 are in normal reference range.
6. Subject has taken any oral, injectable, or IV steroids within 8 weeks from time of screening visit, or plans to take any oral, injectable, or IV steroids during the course of the study
7. Subject is currently abusing illicit drugs
8. Subject is currently abusing prescription drugs
9. Subject is currently abusing alcohol
10. Subject has sickle cell disease or hemoglobinopathy
11. Subject has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening or plans to receive red blood cell transfusion or erythropoietin over the course of study participation
12. Subject diagnosed with current eating disorder such as anorexia or bulimia
13. Subject has been diagnosed with chronic kidney disease that results in chronic anemia
14. Subject is on dialysis

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2013-11-26 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Lee, MD, Study Director — Medtronic Diabetes
Locations (43):
- United States (43):
  - Medical Investigations, Inc., Little Rock, Arkansas
  - AMCR Institute, Escondido, California
  - Valley Research, Fresno, California
  - Center of Excellence in Diabetes & Endocrinology, Sacramento, California
  - So Cal Diabetes, Torrance, California
  - Barbara Davis Center (1), Aurora, Colorado
  - Barbara Davis Center (2), Aurora, Colorado
  - East Coast Institute for Research, Jacksonville, Florida
  - Endocrine Associates of Florida, P.A., Lake Mary, Florida
  - TLC Diabetes Healthcare Consultants & Education Inc., Naples, Florida
  - Pediatric Endocrine Associates, Tampa, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - East Alabama Endocrinology PC, Columbus, Georgia
  - Endocrine Research Solutions, Roswell, Georgia
  - The University of Chicago, Chicago, Illinois
  - Isaiah Pittman IV, MD, Terre Haute, Indiana
  - Good Samaritan Hospital Physician Services, Vincennes, Indiana
  - Iowa Diabetes and Endocrinology Center, Des Moines, Iowa
  - Imperial Health, Lake Charles, Louisiana
  - Eastern Shore Diabetes and Endocrinology Center, Salisbury, Maryland
  - University of Michigan Diabetes Research Center, Ann Arbor, Michigan
  - Grunberger Diabetes Institute, Bloomfield Hills, Michigan
  - Spectrum Health System, Grand Rapids, Michigan
  - International Diabetes Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - The Diabetes Center, Ocean Springs, Mississippi
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Billings Clinic, Billings, Montana
  - Glacier View Research Institute-Endocrinology, Kalispell, Montana
  - Complete Endocrinology, Lincoln, Nebraska
  - Diabetes, Endocrinology, Metabolism Specialties, Teaneck, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Rochester General Hospital, Rochester, New York
  - Joslin Diabetes Center, Syracuse, New York
  - University at Buffalo, The State University of New York, Williamsville, New York
  - Physicians East, PA, Greenville, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - AM Diabetes and Endocrinology Center, Bartlett, Tennessee
  - Endeavor Clinical Trials, San Antonio, Texas
  - Consano Clinical Research, LLC, San Antonio, Texas
  - Northeast Clinical Research of San Antonio, LLC, Schertz, Texas
  - Southwestern Vermont Health Care, Bennington, Vermont
  - Tri-Cities Diabetes and Endocrinology Center, Richland, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Medtronic MiniMed 530G Insulin Pump: All subjects received diabetes treatment using the Medtronic MiniMed 530G insulin pump.
  Medtronic MiniMed 530G Insulin Pump
Period: Overall Study
Arm/Group | Medtronic MiniMed 530G Insulin Pump
Started | 372
Completed | 305
Not Completed | 67
Not completed — Death | 3
Not completed — Lost to Follow-up | 12
Not completed — Withdrawal by Subject | 52

BASELINE CHARACTERISTICS:
Arm/Group | Medtronic MiniMed 530G Insulin Pump
Number analyzed (Participants) | 372
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.5 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201
  Male | 171
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 351
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 372

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in A1C From Baseline to 1 Year
Description: Comparison of A1C measurement from baseline to end of study in the CEP266 study population.
  The overall mean change in A1C from baseline will be estimated and compared by a non-inferiority test with an A1C margin of 0.4% and a significance level of 0.025 (one-sided) with the CEP 266 study population.
Time Frame: 1 year
Population: Among the 372 enrolled subjects, 298 had both baseline and end of study A1c.
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Medtronic MiniMed 530G Insulin Pump
Number analyzed (Participants) | 298
percentage | 0.034 [-0.03 to 0.098]
Statistical Analysis 1: Comparison: Medtronic MiniMed 530G Insulin Pump; Test type: Non-Inferiority — non-inferiority test with an A1C margin of 0.4% and a significance level of 0.025 (one-sided); Mean Difference (Net) = 0.034, 95% CI 2-sided [-0.03 to 0.098]

2. Secondary Outcome: Mean Change in A1C From Baseline to 1 Year, Baseline A1c Below 7%
Description: Mean Change in A1C From Baseline to 1 Year, for subjects with baseline A1c below 7%.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Medtronic MiniMed 530G Insulin Pump
Number analyzed (Participants) | 83
percentage | 0.32 (0.53)

3. Secondary Outcome: Mean Change in A1C From Baseline to 1 Year, Baseline A1c of 7% to 9%
Description: Mean Change in A1C From Baseline to 1 Year, for subjects with Baseline A1c of 7% to 9%
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Medtronic MiniMed 530G Insulin Pump
Number analyzed (Participants) | 187
percentage | -0.04 (0.67)

4. Secondary Outcome: Mean Change in A1C From Baseline to 1 Year, Baseline A1c > 9%
Description: Mean Change in A1C From Baseline to 1 year, for subjects with Baseline A1c > 9%
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Medtronic MiniMed 530G Insulin Pump
Number analyzed (Participants) | 28
percentage | -0.39 (0.96)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Medtronic MiniMed 530G Insulin Pump
All-Cause Mortality (participants affected / at risk) | 3/372
Serious Adverse Events (participants affected / at risk) | 19/372
Other Adverse Events (participants affected / at risk) | 37/372
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medtronic MiniMed 530G Insulin Pump (N=372)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 1 (1)
Chest pain (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 5 (5)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Mixed hepatocellular cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (4)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medtronic MiniMed 530G Insulin Pump (N=372)
Abscess limb (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (3)
Convulsion (Nervous system disorders) | 1 (1)
Dermatophytosis (Infections and infestations) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (13)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (4)
Infusion site erythema (General disorders) | 1 (1)
Infusion site infection (Infections and infestations) | 1 (1)
Ketonuria (Renal and urinary disorders) | 1 (1)
Medical device site reaction (General disorders) | 1 (1)
Nerve injury (Injury, poisoning and procedural complications) | 1 (1)
Puncture site haemorrhage (General disorders) | 9 (14)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Scar (Injury, poisoning and procedural complications) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT02003898/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT02003898/SAP_001.pdf